CLINICAL TRIAL: NCT06068374
Title: Acute Effects of Breaks From Sedentary Behavior With Dual Tasks on Cerebral Blood Flow, Cognitive Function, Blood Pressure and Vascular Function in the Elderly
Brief Title: Breaks From Sedentary Behavior With Dual Tasks in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Raphael Mendes Ritti Dias, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Break_Elderly
Record Dates: First submitted 2023-09-22; First posted 2023-10-05 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Aging
Keywords: sedentary behavior; physical activity; cognitive function; vascular function
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The evaluator of flow-mediated dilation is blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Break dual task (Experimental): Subjects will remain seated for three hours; however, every 30 minutes the subjects will be instructed to stand and take short walks with low intensity and perform a cognitive task
  Interventions: Other: Break of sedentary behavior with dual task
- Standard break (Active Comparator): Subjects will remain seated for three hours, however, every 30 minutes the subjects will be instructed to stand and take short walks at low intensity for two minutes,
  Interventions: Other: Break of sedentary behavior with walking
- Control session (No Intervention): Subjects will remain seated for three hours

INTERVENTIONS:
Other: Break of sedentary behavior with dual task — Patients will interrupt sedentary behavior performing walking and cognitive activities simultaneously
  Arms: Break dual task
Other: Break of sedentary behavior with walking — Patients will interrupt sedentary behavior performing walking
  Arms: Standard break

SUMMARY:
The aim of this project will be to compare the acute effects of breaks from sedentary behavior using dual-tasking on cerebral blood flow, vascular function, cognitive functions and blood pressure in elderly people. Participants will perform, in random order, three experimental sessions (control, break with dual-task and standard break ([walk]). All sessions will have a period of 4 hours in sedentary behavior. In the standard break session and in the break session with dual-task participants will take walking and dual-task breaks every 30 minutes, and in the control session they will remain seated without breaks. Before and after this period, cerebral blood flow, vascular function, cognitive functions and blood pressure will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years or over
* be physically independent based on the Katz Test
* have no history of heart attack
* not having suffered a stroke
* not have heart failure
* do not have joint problems that prevent them from carrying out experimental sessions
* do not have a history of neurodegenerative diseases
* obtain ≥ 26 points in the Montreal Cognitive Assessment (MoCA)
* are not involved in the practice of regular, systematic physical activity more than once a week over the last six months prior to the start of the study
* not be smokers and morbidly obese.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Cerebral blood velocity [centimeters per second] | Before and 20 minutes after the intervention for 5 minutes
  Mean arterial velocity of middle cerebral artery will be measured using a transcranial doppler
Cognitive function - The Trail Making Tests [seconds] | Before and 30 minutes after the intervention
  The Trail Making Tests (A and B) will be used to assess executive function and attention. Part A will determine psychomotor speed and require the participant to draw lines connecting sequentially circled numbers, such as drawing a line from 1 to 2, 2 to 3, and 3 to 4. Part B will consist of circled numbers and letters. Participants will be instructed to draw a line as quickly and as accurately as possible from 1 to A, A to 2, 2 to B, B to 3, and so on, until they complete the task. The time in seconds will be recorded in seconds after the end of each stage. After carrying out the tests, the differences between the completion times for part B - A will be calculated.
Cognitive function - Stroop test [seconds] | Before and 32 minutes after the intervention
  A computerized version of the Stroop test will be used in this study, using the Testinpacs® program. The tasks will be viewed on a notebook screen approximately 90 cm away from the participant. Answers to a set of tasks will be given as quickly as possible via two buttons. The cognitive portion of the Stroop test will be used as a psychometric test to assess cognition, being related to the executive functions of decision-making and inhibitory control exercised by the prefrontal cortex. The capacity for selective attention and response control will be estimated as the time difference between the third condition and the second condition. Smaller differences will indicate better selective attention and conflict resolution.
Cognitive function - verbal fluency [number of animal names reported] | Before and 35 minutes after the intervention
  The task will consist of recalling words that begin with the letter "F", for 60 seconds. The final score will be determined according to the number of correct words reported in 60 seconds. In the semantic modality, participants must evoke as many animals as possible in 60 seconds. The final score will be determined according to the number of animal names reported in 60 seconds.

SECONDARY OUTCOMES:
Resting systolic and diastolic blood pressures [mmHg] | Before and 10 minutes after the intervention
  Resting systolic and diastolic blood pressures will be assessed with an automatic blood pressure monitor (HEM-742, Omron Healthcare, Japan).
Resting heart rate [bpm] | Before and 10 minutes after the intervention
  Resting heart rate will be assessed with an automatic blood pressure monitor (HEM-742, Omron Healthcare, Japan).
Ambulatory systolic, diastolic, and mean blood pressures monitoring [mmHg] | 45 minutes after the intervention
  The systolic, diastolic, and mean blood pressures during 24 hours will be measured using a non-invasive oscillometric device (Dynamapa)
Vascular function [%] | Before and 10 minutes after the intervention
  Vascular function will be measured with the flow-mediated dilation according to the global recommendations on popliteal artery before and after 15 minutes of intervention by a bidimensional ultrasonography device with spectral Doppler and linear transducer.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Dias, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: One year after the completion
Access Criteria: Upon request